CLINICAL TRIAL: NCT05218473
Title: Using 14-day Continuous Electrocardiography Patch Monitoring to Detect Paroxysmal Atrial Fibrillation in Patients With Acute Ischemic Stroke: a Protocol for a Prospective Single-arm Study Using a Historical Control for Comparison
Brief Title: Using 14-day Continuous Electrocardiography Patch Monitoring to Detect Paroxysmal Atrial Fibrillation After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jiann-Der Lee, Associate Clinical Professor, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202101821B0C601
Record Dates: First submitted 2022-01-06; First posted 2022-02-01 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation; Ischemic Stroke
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This is an interventional study without concurrent controls. We will compare the detection rate of paroxysmal atrial fibrillation in acute ischemic stroke patients without known atrial fibrillation, using 14-day continuous ECG patch monitoring, with a historical control group of patients who received serial 12-lead ECGs or 24-hour Holter monitoring.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged ECG monitoring group (Experimental): Patients receive 14-day continuous electrocardiography patch monitoring
  Interventions: Diagnostic Test: Prolonged ECG monitoring
- Conventional procedure group (Active Comparator): Patients received serial 12-lead electrocardiograms once daily for five days or 24-hour Holter monitoring
  Interventions: Diagnostic Test: Conventional procedure group

INTERVENTIONS:
Diagnostic Test: Prolonged ECG monitoring — Using 14-day continuous electrocardiography patch monitoring to increase the detection rate of paroxysmal atrial fibrillation in acute ischemic stroke patients without known atrial fibrillation.
  Arms: Prolonged ECG monitoring group
Diagnostic Test: Conventional procedure group — Using serial 12-lead electrocardiograms once daily for five days or conventional 24-h Holter monitoring to detect new atrial fibrillation
  Arms: Conventional procedure group

SUMMARY:
In this prospective, single-center, open-label, non-randomized, single- arm, historically controlled study, we will compare the detection rate of paroxysmal atrial fibrillation in acute ischemic stroke patients without known atrial fibrillation, using 14-day continuous electrocardiography patch monitoring, with a historical control group of patients who received serial 12-lead electrocardiograms once daily for five days or conventional 24-hour Holter monitoring. The study will be conducted in Chang Gung Memorial Hospital at Chiayi, Taiwan, from February 2022 to December 2024.

DETAILED DESCRIPTION:
Study design In this prospective, single-center, open-label, non-randomized, single- arm, historically controlled study, we will compare the detection rate of paroxysmal atrial fibrillation in acute ischemic stroke patients without known atrial fibrillation, using 14-day continuous ECG patch monitoring, with a historical control group of patients who received serial 12-lead ECGs or 24-hour Holter monitoring. The study will be conducted in Chang Gung Memorial Hospital at Chiayi, Taiwan, from February 2022 to December 2024.

Study population Patients are eligible to participate if they meet the inclusion criteria and without the exclusion criteria. A historical control group will be drawn from our randomized clinical trial, which have been executed between October 2015 and October 2018, and aimed to evaluate the detection rate of new atrial fibrillation in acute ischemic stroke patients without known atrial fibrillation. Patients in the historical control group will have received serial 12-lead ECGs once daily for five days or conventional 24-hour Holter monitoring. In this study, serial ECGs had comparable detection rate of paroxysmal atrial fibrillation compared with 24-hour Holter monitoring. All clinical information and outcomes have been prospectively recorded.

Trial intervention Eligible patients in this study will receive 14-day continuous ECG patch monitoring.

A 14-day ECG patch monitor (EZYPRO, UG02, Sigknow Biomedical Co., Ltd, Taipei, Taiwan) was developed and evaluated in this study. The EZYPRO is a lightweight, waterproof, single-lead ECG device with no external leads or wires and allows for continuous ECG monitoring for up to 14 days. The data were collected and recorded by the investigators and analyzed with the proprietary analytical software and qualified ECG technicians from Sigknow Biomedical Co., Ltd. and adjudicated by attending cardiologists at the study site.

Study outcomes The primary outcome will be the percentage of patients with new atrial fibrillation. Atrial fibrillation was defined as an episode of irregular heart rhythm, without detectable P waves, lasting more than 30 seconds.

Sample size We calculated sample size based on our preliminary data preceding the actual conduct of this trial. New AF was detected in 7.6% of acute ischemic stroke patients who received serial ECG or Holter monitoring. Studies with monitoring lasting ≥ 7 days have been shown to detect AF in 15% of patients after ischemic stroke or transient ischemic attack. The total sample sizes will be 120 for the long-term monitoring group and 120 for the control group. The estimated detection rate of new AF is 7.6% for the control group and 20% for the long-term monitoring group, with 80% power and a two-sided α of 0.05. To allow for dropouts, 150 patients would be recruited in long-term monitoring group.

Statistical analysis Statistical analyses will be performed using the SPSS statistical software (V.25). The Kolmogorov-Smirnov test will be used to examine the normality of continuous variables. The Mann-Whitney U test and Student's t-test will be used to test for differences between the two groups, as appropriate. Categorical data will be analyzed using the χ2 test. A propensity score matching analysis will be used to measure and balance predetermined covariates between two groups. A logistic regression model will be used to test independent variables for the measured outcomes. Variables showing a p value of < 0.1 for univariate analysis will be entered into the multivariate logistic analysis using the forward selection method. All tests will be two-tailed, and a p value of < 0.05 is considered to indicate a statistically significant difference.

ELIGIBILITY:
Inclusion criteria

* Acute ischemic stroke defined as an acute episode of neurological dysfunction caused by focal cerebral infarction and/or a corresponding lesion on brain imaging
* Stroke symptoms within 7 days
* Age ≥ 50 years
* At least one 12-lead ECG has already been obtained as part of the routine clinical workup after admisison, and no ECGs have shown any episodes of atrial fibrillation or atrial flutter

Exclusion criteria

* History of atrial ﬁbrillation/atrial flutter or documented atrial ﬁbrillation/atrial flutter prior to enrollment
* Intracerebral hemorrhage in medical history
* Implanted pacemaker device or cardioverter/deﬁbrillator
* End stage renal disease
* Endocarditis
* Untreated hyperthyroidism
* Myocardial infarction or cardiac surgery less than one month prior to index stroke
* Any finding on echocardiography for which there is already an evidence-based indication for long-term anticoagulation (e.g. mechanical heart valve, thrombus, etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-21 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Paroxysmal atrial fibrillation | day 14
  The detection rate (%, percent) of new paroxysmal atrial fibrillation in each arm